CLINICAL TRIAL: NCT04901559
Title: Subjective Outcomes After ACL Reconstruction With BQT Autograft
Status: Completed | Type: Observational
Sponsor: Region Zealand (Other)
Responsible Party: Principal Investigator, Jesper Glerup, Medical student, Region Zealand
Other Study IDs: BQT-1
Record Dates: First submitted 2021-05-12; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: ACL Injury; Knee Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BQT: Patients treated with the Bone Quadriceps Tendon (BQT) autograft
  Interventions: Procedure: Graft type at ACLR
- STG: Patients treated with the Semitendinosus-Gracilis (STG) autograft
  Interventions: Procedure: Graft type at ACLR
- BPTB: Patients treated with the Bone-Patellar Tendon-Bone (BPTB) autograft
  Interventions: Procedure: Graft type at ACLR

INTERVENTIONS:
Procedure: Graft type at ACLR — The choice of graft at primary ACL Reconstruction

SUMMARY:
The purpose of the study is to compare short-term patient reported outcome measures (PROM) of Bone-Quadriceps-Tendon (BQT) autograft with Semitendinosus-Gracilis (STG) and Bone-Patellar-Tendon-Bone (BPTB) autografts following Anterior Cruciate Ligament Reconstruction (ACLR).

The PROM used are Knee Injury and Osteoarthrithis Outcome Score (KOOS) and Tegner. Difference in change in KOOS, KOOS subscales and Tegner from preoperative baseline to one-year follow-up and absolute KOOS, KOOS subscales and Tegner at one-year follow-up were evaluated. All of which were BQT compared to STG and BPTB, respectively. The primary outcome is change in KOOS from preoperative baselinge to one-year follow-up. Other outcomes are secondary.

The hypothesis was that patients receiving the BQT autograft show similar results in KOOS, KOOS subscales and Tegner as patients receiving STG or BPTB autografts.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Revision ACL Surgery
* Multiligament surgery
* Nonresponders in PROM at preoperative baseline or one-year follow-up

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the nationwide Danish Knee Ligament Reconstruction Register (DKLR) recruited from both private and public clinics from January 1st 2005 through December 31st 2018.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score from preoperative baseline to one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively

SECONDARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score subscale Pain from preoperative baseline to one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Change in Knee Injury and Osteoarthritis Outcome Score subscale Symptoms from preoperative baseline to one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Change in Knee Injury and Osteoarthritis Outcome Score subscale Activities of Daily Living (ADL) from preoperative baseline to one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Change in Knee Injury and Osteoarthritis Outcome Score subscale Sports/Recreation from preoperative baseline to one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Change in Knee Injury and Osteoarthritis Outcome Score subscale Quality of Life (QoL) from preoperative baseline to one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Change in Tegner activity score from preoperative baseline to one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Absolute results of Knee Injury and Osteoarthritis Outcome Score subscale Pain at one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Absolute results of Knee Injury and Osteoarthritis Outcome Score subscale Symptoms at one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Absolute results of Knee Injury and Osteoarthritis Outcome Score subscale Activities of Daily Living (ADL) at one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Absolute results of Knee Injury and Osteoarthritis Outcome Score subscale Sports/Recreation at one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Absolute results of Knee Injury and Osteoarthritis Outcome Score subscale Quality of Life (QoL) at one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively
Absolute results of Tegner activity score at one-year follow-up | 1 year
  BQT compared to STG and BPTB, respectively

IPD SHARING:
Plan to Share IPD: No